CLINICAL TRIAL: NCT00368732
Title: Gene and Nutrient Etiologies of Human Heart Defects
Brief Title: Genetic and Nutritional Causes of Heart Birth Defects
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Gary M. Shaw, DrPH, California Birth Defects Monitoring Program
Other Study IDs: 1352; R01HL085859 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2007-12

CONDITIONS: Heart Defects, Congenital
Keywords: Congenital Heart Defects
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Buccal cell collection

SUMMARY:
Each year in the United States, thousands of babies are born with heart defects. Women who take folic acid during pregnancy have a lower risk of giving birth to infants with heart defects, but the reason for this remains unknown. This study will examine the relationship between genes, nutrition, and the occurrence of heart defects in infants.

DETAILED DESCRIPTION:
Congenital heart defects are the most common type of birth defect; each year, more than 30,000 babies in the United States are born with this kind of abnormality. Conotruncal heart defects, considered to be a very serious type of defect, involve a structural abnormality in the chambers of the heart or blood vessels that lead to and from the heart. Infants born with conotruncal defects must undergo complex open heart surgery, and there is a high fatality rate. Folic acid supplementation during pregnancy has been shown to reduce the risk of conotruncal defects. However, some women who take folic acid during pregnancy still give birth to infants with conotruncal defects. Specific genes may influence the way individuals metabolize folic acid, and variations in these genes may make some infants more prone to developing heart defects. This study will examine the relationship between genes, maternal nutritional intake, and conotruncal heart defects. The results from this study may help to determine genetic and nutritional causes of congenital heart defects.

This study will use previously collected data on 550 infants born with conotruncal defects and 1060 infants born without heart defects. There will be no study visits specifically for this study. Infant DNA will be analyzed for genes that may play a role in folate metabolic pathways. Blood previously collected from the mothers during pregnancy will be analyzed for differences in nutrient intake. Specifically, levels of folic acid, choline, vitamin B12, and methionine will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Conotruncal heart defect

Exclusion Criteria:

* If part of control group, must not have heart defect

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mothers of babies with heart defects and mothers of babies without any malformation.
Sampling Method: Probability Sample
Enrollment: 1610 (Actual)
Dates: Start 2006-07; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary M. Shaw, DrPH, Principal Investigator — California Birth Defects Monitoring Program
Locations (1):
- California Birth Defects Monitoring Program, Berkeley, California, United States

REFERENCES:
- See also: Click here for the California Birth Defects Monitoring Program web site — http://www.cbdmp.org